CLINICAL TRIAL: NCT04342728
Title: Coronavirus Disease 2019- Using Ascorbic Acid and Zinc Supplementation (COVIDAtoZ) Research Study A Randomized, Open Label Single Center Study
Brief Title: Coronavirus 2019 (COVID-19)- Using Ascorbic Acid and Zinc Supplementation
Acronym: COVIDAtoZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Milind Desai, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 20-361
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: COVID; Corona Virus Infection
Keywords: COVID-19; Viral Infection; Infection; Coronavirus-19; Ascorbic Acid; Zinc Gluconate
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Virus Diseases; Infections | interventions — Ascorbic Acid; gluconic acid; Zinc; Standard of Care

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, open label four arm study (1. Zinc only 2. Zinc and ascorbic acid 3. Ascorbic acid only 4. Standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ascorbic Acid (Active Comparator): 8000 mg of ascorbic acid divided into 2-3 doses/day with food.
  Interventions: Dietary Supplement: Ascorbic Acid
- Zinc Gluconate (Active Comparator): 50 mg of zinc gluconate to be taken daily at bedtime
  Interventions: Dietary Supplement: Zinc Gluconate
- Ascorbic Acid and Zinc Gluconate (Active Comparator): 8000 mg of ascorbic acid divided into 2-3 doses/day with food and 50 mg of zinc gluconate to be taken daily at bedtime.
  Interventions: Dietary Supplement: Ascorbic Acid and Zinc Gluconate
- Standard of Care (Other): Standard of care medications only as prescribed by patient's physician.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Ascorbic Acid — Readily available marketed open label ascorbic acid
  Other Names: Vitamin C
  Arms: Ascorbic Acid
Dietary Supplement: Zinc Gluconate — Readily available marketed open label zinc gluconate
  Other Names: Zinc
  Arms: Zinc Gluconate
Dietary Supplement: Ascorbic Acid and Zinc Gluconate — Readily available marketed open label ascorbic acid and zinc gluconate
  Other Names: Vitamin C and Zinc
  Arms: Ascorbic Acid and Zinc Gluconate
Other: Standard of Care — Readily available prescribed medications/ supplements- None study supplements
  Other Names: Standard prescribed medications/ supplements
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to examine the impact of ascorbic acid (vitamin c) and zinc gluconate in reducing duration of symptoms in patients diagnosed with coronavirus disease 2019 (COVID-19). Patients above the age of 18 who present to the Cleveland Clinic outpatient testing and receive a positive test for COVID-19 will be invited to participate.

DETAILED DESCRIPTION:
We aim to see whether ascorbic acid and zinc gluconate which has limited side effect profile and is readily available over the counter can decrease the duration of symptoms seen in patients with new diagnosis of COVID-2019. A secondary purpose is to see whether Zinc and/or Ascorbic acid supplementation can prevent progression of the severe manifestations of the disease including development of dyspnea and acute respiratory distress syndrome which may require hospitalization, mechanical ventilation, and or lead to death.

This is a single-center, prospective, randomized study which plans to enroll 520 patients with a principal diagnosis of COVID-2019, managed in an outpatient setting, who presented after being sent by a healthcare provider to get tested and receive a PCR (Polymerase Chain Reaction) -assay based confirmed diagnosis of the disease. All patients who agree to participate in the study will answer a baseline questionnaire about their symptoms at the time of inclusion. Patients will then be randomized to one of 4 study arms. Patients in Arm A (n=130) will receive vitamin C (to be taken divided over 2-3 times a day with meals), patients in Arm B (n=130) will receive zinc gluconate to be taken at bedtime, patients in Arm C (n=130) will receive both vitamin C (to be taken divided over 2-3 times a day with meals) and zinc gluconate (taken at bedtime). Patients in arms A, B and C will take study supplements daily for 10 days. Patients in Arm D (n=130) will not receive any of the study medications and continue on standard of care. Patients will then track their symptoms daily from day 0 to day 28 answering 12 basic questions on illness severity.They will stop filling out their daily questions once they reach reach the end of the 28 day study period or at time of hospitalization; whichever comes first . Study team members will call patients at days 7, 14, 21, and 28 of the study period to assess need for hospitalization, ER visit, or additional medications prescribed by a healthcare provider, and any side effects from the supplements that the patient could have experienced.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 18 years presenting to Cleveland Clinic Health System in Ohio and Florida who test positive for COVID-19 having any of the following symptoms

  1. Fever or chills
  2. Shortness of breath or difficulty breathing
  3. Cough
  4. Fatigue
  5. Muscle or body Aches
  6. Headache
  7. New loss of taste
  8. New loss of smell
  9. Congestion or runny nose
  10. Nausea
  11. Vomiting
  12. Diarrhea

Women of child bearing potential:

1. have had a menstrual period within the past 30 days, or
2. have had previous sterilization, or
3. are perimenopausal (less than 1 year) who have a negative pregnancy test, or
4. women of childbearing potential who do not meet the above and have a negative pregnancy test.

Exclusion Criteria:

* Patients who are found to be positive during hospitalization
* Patients who reside outside Ohio or Florida.
* Pregnant women:

  1. Current known pregnancy
  2. Positive pregnancy test (women of child bearing potential who have not had previous sterilization as defined as hysterectomy or tubal ligation)
* Women of childbearing potential who do not meet the above criteria, last menstrual period greater than 30 days and have a positive pregnancy test.
* Lactating Women
* End stage kidney disease
* Advanced liver disease awaiting transplant
* History of Calcium Oxalate kidney stones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Symptom Reduction | 28 days
  Number of days to reach a 50 percent reduction in the cumulative 0-36 symptom score with each symptom evaluated on a 0-3 scale. Assessed symptoms are Fever, Cough, Shortness of Breath, Fatigue, Muscle or body aches, Headache, New loss of taste, New loss of smell, Congestion or runny nose, Nausea, Vomiting, Diarrhea. Each patient will have a composite score ranging from 0-36/day

SECONDARY OUTCOMES:
Symptom Resolution: Fever | 28 days
  The number of days required to reach a score of 0 from the symptom category of fever based on a 0-3 scale: 0 = ≤98.6, 1 = >98.6- 100.6, 2 = > 100.6 - 102.6, 3 = >102.6
Symptom Resolution: Cough | 28 days
  The number of days required to reach a score of 0 from the symptom category of cough based on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe
Symptom Resolution: Shortness of Breath | 28 days
  The number of days required to reach a score of 0 from the symptom category of shortness of breath based on a 0-3 scale: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities
Symptom Resolution: Fatigue | 28 days
  The number of days required to reach a score of 0 from the symptom category of fatigue based on a 0-3 scale: 1=mild fatigue, 2=moderate fatigue, 3=severe fatigue.
Symptom Resolution: Muscle/body aches | 28 days
  The number of days required to reach a score of 0 from the symptom category of muscle/body aches based on a 0-3 scale: 1=mild muscle/body aches, 2=moderate muscle/body aches , 3=severe muscle/body aches.
Symptom Resolution: Headache | 28 days
  The number of days required to reach a score of 0 from the symptom category of headache based on a 0-3 scale: 1=mild headache, 2=moderate headache, 3=severe headache.
Symptom Resolution: New loss of taste | 28 days
  The number of days required to reach a score of 0 from the symptom category of new loss of taste based on a 0-3 scale: 1=mild loss of taste, 2=moderate loss of taste, 3=severe loss of taste.
Symptom Resolution: New loss of smell | 28 days
  The number of days required to reach a score of 0 from the symptom category of new loss of smell based on a 0-3 scale: 1=mild loss of smell, 2=moderate loss of smell, 3=severe loss of smell.
Symptom Resolution: Congestion/ runny nose | 28 days
  The number of days required to reach a score of 0 from the symptom category of congestion/runny nose on a 0-3 scale: 1=mild congestion/runny nose , 2=moderate congestion/runny nose , 3=severe congestion/runny nose .
Symptom Resolution: Nausea | 28 days
  The number of days required to reach a score of 0 from the symptom category of nausea on a 0-3 scale: 1=mild nausea, 2=moderate nausea, 3=severe nausea.
Symptom Resolution: Vomiting | 28 days
  The number of days required to reach a score of 0 from the symptom category of vomiting on a 0-3 scale: 1=mild vomiting, 2=moderate vomiting, 3=severe vomiting.
Symptom Resolution: Diarrhea | 28 days
  The number of days required to reach a score of 0 from the symptom category of diarrhea on a 0-3 scale: 1=mild diarrhea, 2=moderate diarrhea, 3=severe diarrhea.
Day 5 Symptoms | 5 days
  Total symptom composite score at day 5 of study supplementation: Symptom categories of fever based on a 0-3 scale: 0 = ≤98.6, 1 = >98.6- 100.6, 2 = > 100.6 - 102.6, 3 = >102; Cough on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe; Shortness of Breath on a 0-3: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities; and Fatigue on a 0-3 scale: 0 = No fatigue/energetic, 1=mild fatigue, 2=moderate fatigue, 3=severe fatigue.
Hospitalizations | 28 days
  Differences in hospitalization events between the study arms
Severity of Symptoms | 28 days
  Differences in severity of symptoms between study arms
Adjunctive Medications | 28 days
  Differences in number of patients who were prescribed adjunctive medications for their diagnosis between study arms
Supplementation Side Effects | 28 days
  Differences in number of patients in study arms who experienced side effects from the supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, M. D., Principal Investigator — The Cleveland Clinic; Suma Thomas, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD013876. doi: 10.1002/14651858.CD013876.pub3. PMID 36062970
- [Derived] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2021 Jul 22;7(7):CD013876. doi: 10.1002/14651858.CD013876.pub2. PMID 34291813
- [Derived] Thomas S, Patel D, Bittel B, Wolski K, Wang Q, Kumar A, Il'Giovine ZJ, Mehra R, McWilliams C, Nissen SE, Desai MY. Effect of High-Dose Zinc and Ascorbic Acid Supplementation vs Usual Care on Symptom Length and Reduction Among Ambulatory Patients With SARS-CoV-2 Infection: The COVID A to Z Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210369. doi: 10.1001/jamanetworkopen.2021.0369. PMID 33576820